CLINICAL TRIAL: NCT04314141
Title: Surgical and Functional Outcomes, Quality of Life and Patient's Satisfactions Who Have Undergone a Phalloplasty Surgery
Brief Title: Surgical Outcomes, Quality of Life and Patient's Satisfactions With Phalloplasty
Acronym: PHALLO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0759
Record Dates: First submitted 2020-01-02; First posted 2020-03-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Phalloplasty; Surgery
Keywords: phalloplasty; surgery
MeSH Terms: interventions — Quality of Life; Phalloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Transgender patients: Transgender patients who carry out sex reassignment surgery.
  Interventions: Procedure: Evaluation of surgical outcomes, quality of life and patient's satisfactions with phalloplasty
- Cismale patients: Cismale patients who carry out surgery to correct a congenital or acquired lack of penis.
  Interventions: Procedure: Evaluation of surgical outcomes, quality of life and patient's satisfactions with phalloplasty

INTERVENTIONS:
Procedure: Evaluation of surgical outcomes, quality of life and patient's satisfactions with phalloplasty — Send a questionnaire to patients to collect informations about:
  * Sexual quality of life before and after the surgery
  * Satisfaction after surgery
  Data collection in medical file :
  * Surgery outcomes
  * Functional outcomes

SUMMARY:
The phalloplasty is a reconstruction technique, consisting of the neophallus creation.

It is performed in transgender patients in sex reassignment surgery, or in cismale patients to correct a congenital or acquired lack of penis.

There are many surgical techniques, but none is optimal. Surgical and functional outcomes, quality of life and patient's satisfactions with phalloplasty are missing in the international literature.

Urological center of Lyon is a reference center of this kind of surgery and has the possibility to evaluate that.

In this study, 124 transgender and 19 cismale patients with phalloplasty are eligible.

This study will allow us to adapt our practice to the patient's return and improve the information given to patients before their surgery.

It will also improve our surgical techniques, depending on the results achieved.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Patients who have undergone a phalloplasty surgery in the University Lyon Sud Hospital or Croix Rousse Hospital, between 1 January 2007 and 31 October 2018
* Patients with at least one year of back on their surgery procedures
* Transgender patients whose reassignment surgery was validated by a minimum of three members of GRETTIS (Groupe de Recherche, d'Etude et de Traitement des Troubles de l'Identité Sexuelle), including a psychiatrist Or Patients cis males with congenital malformations, or having suffered a total or partial amputation of verge
* Patients who do not oppose orally to participate in the study, after information
* Patients who have given their consent for the audio recording for patients taking part in semi - directive interviews

Exclusion Criteria:

* Minor patients or patients under legal protection
* Refusal to participate in the study
* No understanding of the French language

Ages: 20 Years to 73 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone a phalloplasty surgery in the University Lyon Sud Hospital or Croix Rousse Hospital, between 1 January 2007 and 31 October 2018, with at least one year of back on their surgery procedures.
  Patients concerned with this surgery are :
  * transgender patients whose reassignment surgery was validated by a minimum of three members of GRETTIS, including a psychiatrist.
  * Patients cis males with congenital malformations, or having suffered a total or partial amputation of verge
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
Change of Sexual quality of life of patients with phalloplasty (SEAR questionnaire) from the pre-surgery (Baseline) to one year or more after surgery | One year or more after surgery (baseline)
  Sexual quality of life is evaluated with the SEAR (self esteem and relationship questionnaire), noted in 100.
  It explores different fields of sexual life (sexual report, confidence, self esteem, general relationship with the partner).

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Department, Hospices Civis de Lyon, Pierre-Bénite, France

REFERENCES:
- [Background] Paganelli L, Morel-Journel N, Carnicelli D, Ruffion A, Boucher F, Maucort-Boulch D, Paparel P, Terrier M, Neuville P. Determining the outcomes of urethral construction in phalloplasty. BJU Int. 2023 Mar;131(3):357-366. doi: 10.1111/bju.15915. Epub 2022 Oct 26. PMID 36221955
- [Derived] Pelette R, Morel-Journel N, Carnicelli D, Ruffion A, Paganelli L, Vacheron CH, Terrier M, Madec FX, Neuville P. Functional outcomes after supra-pubic phalloplasty. J Plast Reconstr Aesthet Surg. 2024 Dec;99:263-270. doi: 10.1016/j.bjps.2024.09.065. Epub 2024 Sep 20. PMID 39393169